CLINICAL TRIAL: NCT00068484
Title: A Dose Finding Phase I Trial of the Combination of Topotecan and PS-341, a Novel Proteasome Inhibitor, in Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00044; HIC #12760; R21CA097750 (NIH); CDR0000322889 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Topotecan; trioctyl phosphine oxide; Bortezomib

ARMS (1):
- Treatment (topotecan hydrochloride, bortezomib) (Experimental): Patients receive topotecan IV over 30 minutes on days 1-5. Beginning with course 2, patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: topotecan hydrochloride; Drug: bortezomib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Drugs used in chemotherapy such as topotecan use different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for tumor cell growth. Combining topotecan with bortezomib may kill more tumor cells. This phase I trial is studying the side effects and best dose of topotecan and bortezomib when given together in treating patients with metastatic or unresectable cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of the combination of PS-341 and topotecan. II. Determine the dose limiting toxicities and maximum tolerated dose as well as the recommended phase II doses of the combination.

III. Assess the pharmacokinetics of topotecan alone and in combination with PS-341.

SECONDARY OBJECTIVES:

I. Estimate the objective response rate of a combination of PS-341 and topotecan delivered on days 1-5 every three weeks as defined by the RECIST criteria.

II. Assess the pharmacodynamics of topo I levels. III. Determine the expression of the DNA repair enzyme XRCC1 in tumor biopsies.

OUTLINE: This is a dose-escalation study.

Patients receive topotecan IV over 30 minutes on days 1-5. Beginning with course 2, patients also receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of topotecan and bortezomib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which no more than 1 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A total of 20-25 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective
* Tumor accessible to core needle biopsy and willingness to undergo this procedure prior to the start of treatment
* Evaluable disease as defined in the RECIST criteria
* ECOG performance status =< 2
* Life expectancy of greater than 3 months
* Absolute neutrophil count > 1,500/ul
* Platelets > 100,000/ul
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* Creatinine < 2.0 mg/ml
* Ability to understand and the willingness to sign a written informed consent document
* Metastatic brain or meningeal tumors are allowed if the patient is > 1 month from surgery and/or radiation and is clinically stable with respect to the tumor at the time of the study entry and currently off corticosteroids
* Pregnancy test for pre-menopausal women
* The effects of PS-341 and topotecan on the developing human fetus are unknown; for this reason women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Creatinine clearance < 40 mL/min
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to topotecan, PS-341 or other agents used in this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because topotecan is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with topotecan and PS-341, breastfeeding should be discontinued; these potential risks may also apply to other agents used in this study
* Because patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with topotecan and PS-341 or other agents administered during the study.; appropriate studies will be undertaken for patients receiving combination anti-retroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2003-07; Primary Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities | Up to 3 years
Maximum tolerated dose (MTD) | 21 days

SECONDARY OUTCOMES:
Pharmacokinetics of topotecan hydrochloride | 5 minutes immediately after sample collection
Levels of topoisomerase I | Up to 3 years
DNA repair enzymes | Up to 3 years
Objective response according to the RECIST criteria | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: John Murren, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States